CLINICAL TRIAL: NCT00056940
Title: Randomized Controlled Trial to Prevent Child Violence
Brief Title: Prevention of Violent Behavior Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1R01HD42260-1; 1R01HD042260 (NIH)
Record Dates: First submitted 2003-03-26; First posted 2003-03-27 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Behavior
Keywords: Prevention; Parenting strategies; Media use; Discipline; Firearm storage
MeSH Terms: conditions — Behavior | interventions — Transtheoretical Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Stages of Change
Behavioral: Safety Check approach

SUMMARY:
Violence is one of the major causes of death and injury for children, adolescents, and young adults 10 to 25 years of age. This study will examine the effectiveness of a violence prevention program in pediatricians' offices. The program is designed for families who bring their 2 to 11 year old children in for a well child exam. It focuses on helping parents change behaviors related to the development of violent behavior in children.

DETAILED DESCRIPTION:
More children die violence-related deaths each year than from all natural causes combined. In 2002, the World Health Organization (WHO) reported that 1.6 million people worldwide died from violence in the year 2000; half of these deaths were due to suicides, one-third were due to homicides, and only one-fifth were war related. The United States continues to have the highest number of violence-related deaths of all developed countries.

The WHO has reviewed the effectiveness of worldwide intervention strategies and made recommendations to promote violence prevention throughout the world. Some of the common themes across all countries included: 1) because families play a fundamental role in influencing the propensity for violent behavior, efforts to provide parents with information and strategies for raising nonviolent children are needed; and 2) early interventions to reduce childhood exposure to violence are essential.

In this study, Wake Forest University Health Sciences (WFUHS) and the American Academy of Pediatrics (AAP) will collaborate to evaluate the effectiveness of a pediatric clinician's intervention that has been extensively pilot tested. Pediatric Research in Office Settings (PROS), a program of the AAP, is a national network of practice-based clinicians experienced in research participation. PROS membership consists of more than 697 practices and 1674 clinicians across the country (in 60 AAP Chapters).

This study is being conducted in primary care pediatric clinics across the country that participate in the PROS network.

PROS practices were randomly assigned to either Group 1 (violence prevention intervention) or Group 2 (literacy promotion effort). The study included a total of 137 clinics across the country, 242 practitioners, and 4,890 patients ages 2 to 11 years old. Group 1 providers received a community violence prevention resource worksheet to help them identify community specific assets. Patient families (parent/legal guardian) received tools to help them adhere to provider recommendations. Providers were trained to apply brief techniques of motivational interviewing to help ascertain patient-centered motivation to change violence-related behaviors. Patient families' knowledge, attitudes, and self-reported behaviors were examined prior to the well child exam and at 1 and 6 months after the well child exam. Baseline data were collected in the waiting room; the data forms took 10 minutes to complete. Follow-up telephone interviews were conducted at 1 and 6 months and took 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria

* Parent or legal guardian seen in pediatrician's office for well child exam for their 2 to 11 year old children
* Parent/guardian is with the child the majority of time when the child is at home
* English or Spanish speaking
* Anticipate being at the same phone number for 6 to 12 months

Exclusion Criteria

* Sick child visit
* One child in family already enrolled
* No telephone contact information
* Language other than English or Spanish spoken

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6600
Dates: Start 2001-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
media use time
discipline techniques used
firearm storage patterns

SECONDARY OUTCOMES:
knowledge about appropriate media exposure for children
knowledge about appropriate discipline techniques for children
knowledge about appropriate safe firearm storage

CONTACTS AND LOCATIONS:
Overall Officials: Shari Barkin, MD, MSHS, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt Universitiy School of Medicine, Nashville, Tennessee, United States